CLINICAL TRIAL: NCT06320327
Title: The Effects of Cannabidiol (CBD) Cream on Delayed Onset Muscle Soreness (DOMS and Performance After Exercise
Brief Title: Topical CBD's Effects on Soreness and Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joseph Pastina (Other)
Responsible Party: Sponsor-Investigator, Joseph Pastina, Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 80177
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Muscle Soreness
Keywords: Exercise; Cannabidiol cream
MeSH Terms: conditions — Myalgia; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The research participant's and research personnel conducting the testing will be blinded to who is in the CBD and placebo groups throughout the study. Those in Group 3 (the control group) will be aware that they are in the control group, as they will be skipping the steps involving cream application. The protocols for Group 1 and Group 2 will be identical and the respective cream will be made available to the testers and participants in identical containers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CBD Group (Experimental): This group will apply the CBD cream in accordance with the manufacturer's recommendations at designated time points throughout the study.
  Interventions: Other: Cannabidiol cream
- Placebo Group (Placebo Comparator): This group will apply a placebo moisturizer cream that will match the scent, volume, and viscosity of the CBD cream.
  Interventions: Other: Placebo cream
- Control Group (No Intervention): This group will not apply any cream and will skip all cream-related procedures during the study.

INTERVENTIONS:
Other: Cannabidiol cream — Group 1 will be administered the recommended quantity of CBD cream to be applied at various times throughout the study and used in a specific way instructed by the researcher (the cream is applied via massage through a standardized application method).
  Other Names: Myaderm Advanced RX10 Fast Acting Relief Cream
  Arms: CBD Group
Other: Placebo cream — Group 2 will be administered the recommended quantity of placebo cream to be applied at various times throughout the study and used in a specific way instructed by the researcher (the cream is applied via massage through a standardized application method).
  Other Names: Gold Bond Diabetics' Dry Skin Relief Lotion
  Arms: Placebo Group

SUMMARY:
Exercise-induced muscle damage (EIMD) results from unaccustomed exercise and can lead to delayed onset muscle soreness (DOMS). Impairments associated with EIMD and DOMS can result in moderate-to-severe discomfort and hindered performance. Recently, a compound derived from the cannabis plant, cannabidiol (CBD), has been used as a recovery tool for EIMD and DOMS. Despite the rising popularity of CBD products, their effectiveness in mitigating EIMD and DOMS is unknown. Specifically, to the investigators' knowledge, no clinical trials have been completed to assess the effects of topical CBD cream application on soreness, recovery and performance.

Therefore, the purpose of the present study was to investigate the effects of CBD cream on DOMS and performance after an intensive lower-body exercise protocol. Specifically, the study's aims were:

Aim 1: To assess the effect of topical CBD cream administration on muscle soreness following fatiguing exercise.

Hypothesis 1: CBD cream would decrease perceived muscle soreness when compared to a placebo or control (no cream) group.

Aim 2: To assess the effect of topical CBD cream administration on muscular performance following fatiguing exercise.

Hypothesis 2: Recovery of muscular power would be quicker when CBD cream is applied, compared to a placebo or control (no cream) group.

Aim 3: To assess if topical CBD cream has a localized (if any) or systemic effect on muscle soreness.

Hypothesis 3: Improvements in muscle soreness would only be observed in localized muscles around where the CBD cream was applied.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled experiment examining if CBD cream impacts recovery after exercise. It will be investigated whether or not the potential effects of CBD cream are localized or systemic within the lower body muscles (quadriceps and hamstrings). Furthermore, the study will examine if these potential effects on recovery impact the expected decrements on lower body performance in the days following an intense exercise bout. Overall, the main objective is to determine whether or not CBD cream is an effective recovery method for those who are experiencing DOMS.

Participants will be recruited from volunteers who reside in the Lexington area. Those who participate within the study will be randomly placed into one of three groups by the PI, Dr. Stuart Best: a group that will apply the CBD cream (Group 1), a group that will apply the placebo moisturizer cream (Group 2), or a control group that does not participate in any cream-related procedures (Group 3).

The research participants and research personnel conducting the testing will be blinded to who is in the CBD and placebo groups throughout the study. Furthermore, the PI, who will not participate in any form of testing, will also be responsible for the storage and distribution of the CBD and placebo creams during the study. Those in Group 3 (the control group) will be aware that they are in the control group, as they will be skipping the steps involving cream application. The protocols for Group 1 and Group 2 will be identical and the respective cream will be made available to the testers and participants in identical containers.

A summary of the participant groups is shown below:

Group 1 - CBD Group; This group will apply the CBD cream in accordance with the manufacturer's recommendations throughout the study. Application procedures are described in a section below.

Group 2 - Placebo Group; This group will apply a placebo moisturizer cream that will match the scent, volume, and viscosity of the CBD cream. Application procedures are described in a section below..

Group 3 - Control Group; This group will not apply any cream and will skip all cream-related procedures during the study. During the time that would be designated for cream-related procedures, the control group will rest; this rest period will match the durations of the cream-related procedures for Groups 1 and 2 to keep the delivery of procedures as controlled as possible between groups.

Participants will complete five sessions over the span of 7-11 days. Sessions 1 and 2 will be separated by 3-7 days to wash-out any potential soreness from baseline testing, and Sessions 2-5 will be separated by 24-hr each. A session outline is described below:

Session 1: Anthropometric data, baseline measurements for isokinetic peak torque (PT) and countermovement jump (CMJ) as well as familiarization with the pressure-pain threshold (PPT) test are established. Prior to baseline testing, familiarization with the CMJ and PT instruments and procedures are included during this introductory session.

Session 2 (3-7 days after Session 1): The time between Sessions 1 and 2 ensured each participant began the Session 2 without any residual muscle damage or soreness from Session 1. Participants will complete a digital questionnaire to monitor and evaluate soreness and recovery. Questionnaires will be administered using Research Electronic Data Capture (REDCap) on the investigator's personal computer. Participants will then complete a PPT test, which will serve as their baseline measurement, followed by a fatiguing exercise protocol (FP) designed to induce muscle damage and soreness. The FP consists of repeated maximal effort concentric and eccentric muscle actions at the knee joint (5 sets, 10 reps, 30 seconds rest for both concentric/eccentric knee extension/flexion and eccentric/concentric knee extension/flexion, respectively). A Post-FP questionnaire will be completed to monitor changes in muscle soreness after the FP, followed by the cream application/sitting rest procedures (C/R) for each participant's respective group. The session concludes with a questionnaire (Post C/R) to evaluate the effects of cream/rest, another PPT, and a CMJ assessment.

Session 3 and 4 (24- and 48-hr after Session 2): Sessions 3 and 4 will utilize identical procedures. Participants will complete a Pre-Session questionnaire to monitor soreness and recovery. Then, PPT and CMJ tests are completed. Participants then apply cream or have seated rest according to the respective protocol for their group. After the cream application/sitting procedure occur, participants complete a follow-up Post C/R questionnaire. Lastly, PPT and CMJ are completed again by the participant.

Session 5 (72-hr after Session 2): Session 5 repeats the research procedures of Session 1, with the exclusion of anthropometric testing. To complete Session 5, as well as their participation in the study, each participant will complete a Post-Study questionnaire

Application Procedures:

Cream application procedures will be the same for both CBD and placebo groups, with only the type of cream applied differing between the two groups. Participants will have their quadriceps marked to represent a 'cream application zone'. Similar to the quadriceps PPT, the markings made on the midline of the anterior leg midway between the anterior superior iliac spine (ASIS) and the superior border of the patella will be utilized. However, two new markings will be created to serve as a superior and inferior site: 1) being one-third of the distance between the ASIS and the superior border of the patella; and, 2) two-thirds of the distance between the ASIS and the superior border of the patella. Each participant will first apply the cream to the most superior site on the dominant leg in a clockwise rhythm at a standardized cadence (50 beats·min^-1) for 30 seconds. The participant will then be instructed to proceed inferiorly until all three sites are completed. For each site, participants will be instructed to apply approximately one-third of the total quantity of cream per container. At the conclusion of this process, participants will be told to finish applying any residual cream remaining in the containers across the entire area of cream application. To assess the localized vs systemic effects of CBD cream, cream will only be applied to the quadriceps in both the CBD and placebo groups. Participants within the control group will be instructed to sit in a relaxed position for 3 minutes. This duration has been chosen because it matches the total time of the cream application for CBD and placebo groups.

ELIGIBILITY:
Inclusion Criteria:

* Physically healthy
* Age 18-45
* Available for 5 sessions over the span of 2 weeks
* Untrained (have not been participating in a structured resistance training routine for the past 2 months that includes 2 days of lower body resistance training per week)

Exclusion Criteria:

* Have not suffered a lower body injury in the previous 3 months
* Be allergic to any ingredients within the CBD or placebo creams (ingredients listed in informed consent form)
* Be pregnant

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Vertical Jump Test | Baseline and immediately post exercise, then 24, 48, and 72 hours post-exercise (pre- and post-cream/rest).
  The vertical jump, or countermovement jump (CMJ), test will utilize the ForceDecks Dual Force Plate System by Vald Performance to measure peak force production and vertical jump height (one plate for each leg; sampling frequency = 1,000 Hz).

SECONDARY OUTCOMES:
Peak Isokinetic Torque Test | Baseline and Session 5 (72 hours post-exercise)
  The Peak Isokinetic Torque Test will use the Biodex, an isokinetic dynamometer to establish measures for concentric and eccentric peak isokinetic torque during knee extension and knee flexion.This test requires a maximal effort on 5 repetitions, and the highest isokinetic torque value of the five repetitions will be documented.
Pressure-Pain Threshold Test | Baseline and immediately post exercise, then 24, 48, and 72 hours post-exercise (pre- and post-cream/rest).
  The pressure-pain threshold test (PPT) is designed to provide a quantitative measure of muscular sensitivity. It will be used to provide a subjective measure of soreness. The test utilizes a compact digital algometer equipped with a 1-cm2 rubber tip that, when pressed against a surface, will provide a pressure reading as force is applied to a surface. The reading will be provided in Newtons (N) and converted to kilopascals (kPa) for analysis (1 N/cm2 = 10 kPa). For the PPT, the subject will have four markings (indicated below) and pressure will be applied to each marking using the algometer using a standardized method. The subject will indicate discomfort rather than pressure, and that value will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart A Best, PhD, Principal Investigator — University of Kentucky
Locations (2):
- United States (2):
  - Seaton Center Building, Lexington, Kentucky
  - Multidisciplinary Science Building, Lexington, Kentucky

DOCUMENTS (1):
  • Informed Consent Form (2022-08-04): https://cdn.clinicaltrials.gov/large-docs/27/NCT06320327/ICF_000.pdf